CLINICAL TRIAL: NCT01857635
Title: Use of TpCO2 (Transcutaneous CO2 Measurement)as PaCO2 Predictor During Non Invasive Ventilation (NIV) in Case of Acute Hypercapnic Respiratory Failure
Brief Title: Use of TpCO2 (Transcutaneous CO2 Measurement) as PaCO2 Predictor During NIV in Case of Acute Hypercapnic Respiratory Failure
Acronym: TpCO2-NIV
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Prof. Philippe Jolliet, Principal investigator, University of Lausanne Hospitals
Other Study IDs: TpCO2-NIV
Record Dates: First submitted 2013-05-15; First posted 2013-05-20 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Hypercapnic Respiratory Failure
Keywords: Acute respiratory failure; Hypercapnia; Non invasive ventilation; Transcutaneous CO2 measurement
MeSH Terms: conditions — Respiratory Insufficiency; Hypercapnia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In patients suffering from hypercapnic respiratory failure and treated by non invasive ventilation (NIV), the interest of using transcutaneous CO2 measurement to evaluate PaCO2 and PaCO2 variation over time is unknown and will be evaluated in this study. Measurements will be done during one-hour NIV treatments.

ELIGIBILITY:
Inclusion Criteria:

* ICU patient equipped with an arterial line
* NIV treatment prescribed by the clinician in charge
* Hypercapnia defined by PaCO2> 42mmHg

Exclusion Criteria:

* Severe hemodynamic instability
* Severe psychiatric disorders
* Denied consent
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care unit patients equipped with an arterial line and requiring non invasive ventilation because of acute hypercapnic respiratory failure
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Comparison between TpCO2 (transcutaneous non invasive CO2 partial pressure measurement) and PaCO2 (obtained by blood gas analysis) values during NIV treatment. | sixty minutes

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jolliet, Prof, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Intensive care and burn unit, University hospital of Lausanne, Lausanne, Switzerland